CLINICAL TRIAL: NCT02254382
Title: Positive Airway Pressure Therapy Study in Sleep Apnea and Diastolic Heart Failure
Acronym: ParadiseHF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment rates too low
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA130514
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Diastolic Heart Failure
Keywords: diastolic heart failure
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adaptive servo ventilation (ASV) (Experimental): This group will receive ventilation therapy (AutoSet CS, ASV device)
  Interventions: Device: Adaptive servo ventilation (ASV)

INTERVENTIONS:
Device: Adaptive servo ventilation (ASV) — Non-invasive Ventilation used to control central and obstructive sleep apnea.
  Other Names: AutoSet CS

SUMMARY:
This is a multicenter, prospective, randomized clinical trial (pilot study). 20 participants with diastolic heart failure will be assigned to ventilation therapy (AutoSet CS ™ ASV device; therapy group). The trial will run for 6 months, after which change in echocardiographic parameters of diastolic left ventricular function, sleep and quality of life parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms of heart failure according to the ESC guidelines
* Echocardiographic evidence of a preserved systolic left ventricular function (echocardiographic left ventricular ejection fraction > 50%)
* Polysomnographic evidence of at least moderate sleep-disordered breathing: apnea-hypopnea index (AHI) > 15 / h with ≥ 50% central events and with with a central AHI of ≥ 10/h (AHI based on total sleeping time, TST)
* BNP or NT-pro BNP ≥ 300 pg / ml
* NYHA class II or III
* Patient tolerates the ventilation treatment (1h sample ventilation)
* Stable drug therapy in the last 4 weeks prior to randomization (no iv diuretic therapy or increasing the dose of diuretics to ≥ 100%)
* Minimum age of patients of 18 years
* patient willing to undergo study procedures
* signed informed consent

Exclusion Criteria:

* Oxygen saturation (sO2) <92% of the days in peace without O2 therapy, measured baseline (start time) in the pulse oximetry or polysomnography in a cape. BGA (the measurement must be max. Lie back 1 week)
* Patients, who have a risk professional with symptomatic sleep apnea
* Known COPD with FEV1 <70%
* patients with NYHA stadium IV
* Advanced congenital heart defects
* pericardial diseases
* Existing PAP or bi-level therapy (including adaptive servo-ventilation) in the last 3 months
* Acute cardiac event in the last 3 months
* BMI ≥ 35kg / m²
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in Apnea-Hypopnea-Index (AHI) | 6 months

SECONDARY OUTCOMES:
Change in total sleeping time (TST) determined by parameters of polysomnography | 6 months
  Total sleeping time (TST) will be measured in minutes (min).
Change in sleep quality determined by parameters of polysomnography | 6 months
  Sleep Quality will be defined by sleep architecture (time spent in sleep Phase 1,2,3 and REM).
Change in sleep efficacy determined by parameters of polysomnography | 6 months
  Sleep efficacy is defined as TST/total time spent in bed, i.e. sleep/awake periods.
Change of echocardiographic parameter of diastolic left ventricular ejection fraction function E/è | 6 months
  E (mitral inflow velocity) and è (mitral annular early diastolic velocity) are parameters to measure filling of the left ventricle with blood.The E/è Ratio gives an estimation of the filling pressure of the left ventricle.
Change of echocardiographic parameters of diastolic function | 6 months
Change of NYHA stage | 6 months
Change of nocturia | 6 months
Changes of questionnaires: ESS | 6 months
  ESS (Epworth Sleepiness Scale) estimates the sleepiness of a person during daytime.
Changes of questionnaires: MLHFQ | 6 months
  MLHFQ (Minnesota Living with Heart Failure) estimates how much HF impairs the daily life of a patient.
Changes of questionnaires (PHQ9) | 6 months
  PHQ9 (Patient health questionnaire) assesses depression of a patient.
Changes of questionnaires (SF12HSQ) | 6 months
  SF12HSQ (short form health status) assesses physical and mental health status.
Change in NT-pro BNP and BNP | 6 months
  NT-pro BNP and BNP (unit ng/l) are comprehensive protein markers of heart diseases, inflammations and cardiovascular disorders. Outcome: Assessment of heart disease status.
Changes in blood gas analysis | 6 months
Change of galactin-3 | 6 months
Change in 6 minute walk test (MWT) | 6 months
Hospitalisations (reason) | 6 months
  Reasons will be described in the corresponding files: Type of disease: Treatment related or unrelated?
Hospitalisations (cumulative length) | 6 months
  Length of hospitalizations are measured in days (d). Severity of disease.
Change in morning blood pressure | 6 months
Change in morning heart rate | 6 months
Occurrence of Adverse Events (AE) and Serious Adverse Events (SAE) | 6 months
Changes in parameters of cardiac repolarisation (QT(c), TpTe(c) intervals, TpTe/QT ratio) in ECG at rest | 6 months
  Electrocardiogram parameters are being put together to assess the patient's heart function status. Outcome: Number of patients with normal heart function.
Changes in occurrence of ventricular and supraventricular arrhythmias (PSG-ECG) | 6 months
  Parameters are being put together to assess the patient's heart function status. Outcome: Number of patients with arrhythmias.
Analysis of compliance data | 6 months
Changes in spiroergometry data (substudy) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Oldenburg, MD, Principal Investigator — Herz- und Diabeteszentrum NRW, Bad Oeynhausen
Locations (2):
- Germany (2):
  - University Hospital Regensburg, Regensburg, Bavaria
  - Heart and Diabetes Centre, Bad Oeynhausen, North Rhine-Westphalia